CLINICAL TRIAL: NCT01723917
Title: Estrogen Receptor-beta phytoSERMs for Management of Menopause and Age-Associated Memory Decline
Brief Title: Phytoserms for Menopause Symptoms and Age-Associated Memory Decline
Acronym: phytoSERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lon Schneider, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AG033288; R01AG033288 (NIH)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Hot Flashes; Memory Loss
MeSH Terms: conditions — Hot Flashes; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PhytoSERM 50 mg tablet (Experimental): Dietary supplement: PhytoSERM tablet to be taken once per day for 12 weeks
  Interventions: Dietary Supplement: PhytoSERM tablet
- PhytoSERM 100 mg tablet (Experimental): Dietary supplement: PhytoSERM tablet to be taken once per day for 12 weeks
  Interventions: Dietary Supplement: PhytoSERM tablet
- Placebo tablet (Placebo Comparator): Dietary supplement: placebo tablet to be taken once per day for 12 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: PhytoSERM tablet
  Arms: PhytoSERM 100 mg tablet; PhytoSERM 50 mg tablet
Dietary Supplement: placebo
  Arms: Placebo tablet

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a soy based dietary supplement (phytoSERM) for hot flashes and age associated memory loss.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women
* ages 45 - 60 (inclusive)
* must have a vasomotor symptom (e.g., hot flash) and a memory complaint

Exclusion Criteria:

* history of clinically significant stroke
* current evidence or history in past 2 years of epilepsy, seizure, focal brain lesion, head injury with loss of consciousness or any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Known allergy to soy derived products; hypersensitivity to estrogens or progestins

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 12 weeks
  as measured by assessment of AEs, co-morbid events, laboratory measures, symptoms and cognitive performance
efficacy | 12 weeks
  change from baseline in neuropsychological (cognitive, functional) test results
efficacy | 12 weeks
  change from baseline in vasomotor symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Lon S Schneider, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Keck School of Medicine, Los Angeles, California, United States

REFERENCES:
- [Derived] Schneider LS, Hernandez G, Zhao L, Franke AA, Chen YL, Pawluczyk S, Mack WJ, Brinton RD. Safety and feasibility of estrogen receptor-beta targeted phytoSERM formulation for menopausal symptoms: phase 1b/2a randomized clinical trial. Menopause. 2019 Aug;26(8):874-884. doi: 10.1097/GME.0000000000001325. PMID 30889096
- [Derived] Hernandez G, Zhao L, Franke AA, Chen YL, Mack WJ, Brinton RD, Schneider LS. Pharmacokinetics and safety profile of single-dose administration of an estrogen receptor beta-selective phytoestrogenic (phytoSERM) formulation in perimenopausal and postmenopausal women. Menopause. 2018 Feb;25(2):191-196. doi: 10.1097/GME.0000000000000984. PMID 28926513